CLINICAL TRIAL: NCT05213585
Title: Treatment of Ocular Demodex Infestation With Topical Ivermectin Cream 1%
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helm Vision Group (Other)
Responsible Party: Principal Investigator, Craig J. Helm, Physician, Helm Vision Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00044340
Record Dates: First submitted 2022-01-20; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: The Focus of the Study is to Assess the Effectiveness of Topical Ivermectin on Eliminating Eyelash Sleeves

STUDY DESIGN:
Intervention Model Description: The untreated eye will be observed in parallel with the contralateral treated eye.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blind to which eye was treated. This is a single arm study in that only 1 treatment protocol is being tested in one eye and the contralateral eye is being used as the control. Masking of the outcomes assessor is being done to eliminate bias from the treating physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treated eyes (Experimental): All participants will have one eye randomly selected for treatment.
  Interventions: Drug: Ivermectin cream
- Untreated eyes (No Intervention): No treatment will be given to the control eye.

INTERVENTIONS:
Drug: Ivermectin cream — Topical application of ivermectin cream to eyelashes of treatment eye.
  Arms: Treated eyes

SUMMARY:
Patients with Demodex infestation of the eyelids will have the sleeves from both eyes cleaned off with microblepharoexfoliation. Afterwards, one eye will be randomly selected for treatment with topical ivermectin 1% cream. The treatment will be repeated on that eye 2 weeks later. Afterwards, the patients will present monthly for photographs of the eyelashes. The photographs will be reviewed by an ophthalmologist outside of our institution who will be blind to which eye was treated and independently grade the amount of sleeves in each eye. The follow-up will be for 6 months after the second treatment.

DETAILED DESCRIPTION:
Informed Consent Form and Authorization to Use and Disclose Protected Health Information

Sponsor / Study Title:

Helm Vision Group / "Treatment of Ocular Demodex Infestation with Topical Ivermectin Cream"

Principal Investigator:

(Study Doctor) Craig Helm, MD

Telephone:

661-259-3937 (24 Hours)

Address: Helm Vision Group 27420 Tourney Rd. Suite 100 Valencia, CA 91355

Background and Purpose

You are being asked to participate in this research study because you have been informed that you have an overgrowth of the eyelash mite (Demodex folliculorum). We expect to enroll 20 subjects in this study.

Mites are small arthropods. Two of these species of mites are specific to humans and are named Demodex folliculorum and Demodex brevis. Demodex folliculorum lives within human hair follicles, whereas Demodex brevis lives in human sebaceous glands.

It is not clearly understood how people get mites but the older one gets the more likely it is that mites will be present. Demodex mites have been determined to be a source of eye and eyelid problems for people of all ages, including children. Having Demodex overgrowth is not a result of poor hygiene. Normal face washing and even the use of baby shampoo lid scrubs do not kill the mites. Ultimately it is thought that everyone gets them, although not everyone seems to be bothered by them. However, they are a cause of suffering for many people.

The presence of Demodex mites is can cause of chronic eyelid inflammation (blepharitis) as well as styes and chalazia (small lumps or cysts within the eyelid). Symptoms of blepharitis include eyelid irritation, redness and itching. Demodex may also be a cause of dry eye syndrome.

The most commonly accepted treatment for eyelash mites involves the use of tea tree oil along the eyelash margin. This treatment though helpful does not usually result in elimination of the organism and can be very irritating depending upon the concentration of tea tree oil that is used. It is known that tea tree oil concentrations of at least 50% are required to kill the mites. Lower concentrations of tea tree oil are commercially available in eyelid wipes and may help to control the mite population but are insufficient to eradicate them.

The purpose of this study is to evaluate the effectiveness of ivermectin cream 1% in eliminating the presence of Demodex infestation of the eyelash follicles. A secondary goal is to evaluate the effectiveness of ivermectin cream 1% in reducing the symptoms of dry eye if any.

A third goal is to determine if study treatment with ivermectin 1% topical cream decreases the salinity of the tears.

Ivermectin cream is FDA-approved for use in rosacea which is a common skin condition associated with redness that affects the face and upper chest. However, the FDA has not approved the use of ivermectin cream for the use of treating Demodex infestation of the eyelids. Therefore, the use of ivermectin cream in this study is investigational.

What Will Happen During the Study?

The study will randomly select one eye to be treated with anti-Demodex study treatment while the other eye will be designated as a control eye and will not be treated with the study treatment.

Both eyes will have the eyelashes cleaned by microblepharoexfoliation (Blephex©). Blephex© is a treatment that uses a soft rotating foam brush soaked in a cleaning solution to remove the scale build-up along the eyelash margins. This build-up (or "biofilm") can constrict the opening of the oil glands (Meibomian glands) that are most important in lubricating the ocular (eye) surface. The Blephex© treatment also removes the debris left behind by the Demodex mites that encircles the base of the eyelashes which are infested. The Blephex procedure is performed after instilling a drop of anesthetic into the eyes. Each eyelid margin is then treated at the base of the eyelashes and lid margin to remove the scaly buildup along the lid margin and to remove the eyelash debris. The procedure takes less than 10 minutes to perform.

Those eyes randomized to the study treatment group will then have the ivermectin cream 1% applied to the base of the eyelashes, eyelids and surrounding skin. The cream will be left in place for 10 to 15 minutes after which point the excess cream will be wiped from the lashes with a saline soaked gauze pad.

At the initial or "baseline" visit each subject will complete a questionnaire which asks questions regarding dry eye and blepharitis symptoms.

A TearLab® test will be performed to measure the saltiness of your tears. The TearLab® test involves taking a tiny sample of your tears from each eye and using a machine to analyze it and determine the salt content. This is used as a measure of the degree of dryness of your eyes. The test is painless.

Photographs of the eyelashes of all four eyelids will then be taken to document the extent of the mite infestation of the eyelids. Mites often leave debris at the base of eyelashes. This debris is called "cylindrical dandruff" or "sleeves." Next, a Blephex© treatment will be performed to remove all of the debris that the mites leave around the eyelashes. Repeat photographs will then be taken to document the successful removal of the mite debris. Afterwards, subjects will be randomized into either the study treatment group or the control group.

Study Treatment Group: Blephex© and study treatment with ivermectin 1% cream Control Group: Blephex© only.

Subjects in the study treatment group will return 2 weeks later for a second application of ivermectin 1% cream.

Photographs, TearLab® tests and the dry eye questionnaire will be repeated at the 2-week and monthly intervals from the date of study treatment for 6 months.

The study will end after 6 months. At this point the control eye will be treated and both eyes treated if necessary.

Risks, Side Effects, and/or Discomforts

Ivermectin

Ivermectin is a drug that has been in worldwide use since 1981 and has proven to be generally very safe. It is on the World Health Organization's List of Essential Medicines, the safest and most effective medicines needed in a health system.

We are using ivermectin cream to avoid the risks associated with its oral use. However it is important that you are aware of all risks associated with ivermectin.

Although oral ivermectin is considered to be safe, a single case of ivermectin-induced severe hepatitis was reported in Switzerland in 2006 using a single dose of 15 mg.

The use of oral ivermectin has been also associated with the following side effects:

* Fatigue (0.9% of subjects)
* Abdominal pain (0.9%)
* Anorexia (0.9%)
* Constipation (0.9%)
* Diarrhea (1.8%)
* Nausea (1.8%)
* Vomiting (0.9%)
* Dizziness (2.8%)
* Sleepiness (0.9%)
* Vertigo (0.9%)
* Tremors (0.9%)
* Itching (2.8%)
* Rash (0.9%)
* Hives (0.9%)
* Low white blood cell count (3%)
* Elevated liver enzymes (2%)
* Anemia

It has also been reported that ivermectin can increase the effect of warfarin (blood thinners, such as Coumadin) when used together.

The use of ivermectin cream has been associated with:

* Burning
* Itching
* Redness
* Stinging of the skin and eyes.

In this study we will apply the ivermectin cream around the eyelids and leave it in place for 10 to 15 minutes. After this period we will remove the excess cream. In our experience to date we have had subjects experience ocular burning and temporary blurring of vision but no other side effects. The blurring of vision has been temporary and in no case interfered with safe driving.

It is possible to have an allergic reaction of the skin to the ivermectin cream although we have not observed this. Absorption of the ivermectin into the body is assumed to be minimal.

BlephEx© You may feel a tickling sensation during the procedure. The eyelid skin may be somewhat irritated afterwards for an hour or two.

Unforeseen Risks

Since the use of the study treatment is investigational, there may be other risks that are unknown. Additionally, there may be unknown risks to a pregnancy, embryo, or fetus if you or your female partner become pregnant.

Study Expectations

You will be enrolled in the study for a 180-day period. During the study period, you will be asked to refrain from using any other type of medicated pad to clean the eyelids and will not be allowed to use any product containing tea tree oil, including tea tree oil-containing soap on the face. Any prescribed glaucoma drops may be used as there are no anti-Demodex properties known with these medications. Antibiotic drops or steroid drops may be prescribed for other ocular conditions as the need arises and will not exclude you from participation in this study.

Alternatives to Participation

You do not have to be in this study to receive treatment for your condition. Please talk to the study doctor about your options before you decide whether or not you will take part in this study.

New Findings

Any new important information that is discovered during the study and which may influence your willingness to continue participation in the study will be provided to you.

Benefits

You may benefit as a result of your participation in this study. There is, however, no guarantee that you will benefit from your participation in this study. Information learned from the study may help other people in the future.

Compensation for Participation

You will not receive any monetary compensation for your participation in this study.

Confidentiality

Records of your participation in this study will be held confidential except when sharing the information is required by law or as described in this informed consent. The Investigator, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the United States Food and Drug Administration (FDA) and the Institutional Review Board (IRB) will be able to inspect and copy confidential study-related records which identify you by name. This means that absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, you will not be identified.

Compensation for Injury

If you become ill or are injured while you are in the study, get the medical care that you need right away. You should inform the healthcare professional treating you that you are participating in this study. If you tell the study staff that you think you have been injured then they will help you get the care you need.

If you are injured as a result of taking the study drug(s) or from procedures done for the purpose of this study, the sponsor will pay for those medical expenses necessary to treat your injury that are not covered by your medical insurance or any other third-party coverage. By signing and dating this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for mistakes.

To pay medical expenses, the sponsor will need to know some information about you like your name, date of birth, and Medicare Beneficiary Identifier (MBI). This is because the sponsor has to check to see if you receive Medicare and if you do, report the payment it makes to Medicare.

Costs

You will be charged the usual and customary charges for office visits and photography as per the contracted rate with your insurance company. There will be no charge to you for the Blephex treatment or application of the ivermectin cream.

Whom to Contact About this Study

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study, please contact the study doctor at the telephone number listed on the first page of this consent document. If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, and/or concerns or complaints regarding this research study, contact:

• By mail: Study Subject Adviser Advarra IRB 6940 Columbia Gateway Drive, Suite 110 Columbia, MD 21046

* or call toll free: 877-992-4724
* or by email: adviser@advarra.com

Please reference the following number when contacting the Study Subject Adviser: Pro00044340.

Voluntary Participation / Withdrawal

Your decision to participate in this study is voluntary. You may choose to not participate or you may withdraw from the study for any reason without penalty or loss of benefits to which you are otherwise entitled and without any effect on your future medical care. However, please note that the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study.

The study doctor or the sponsor can stop your participation at any time without your consent for the following reasons:

* If it appears to be medically harmful to you;
* If you fail to follow directions for participating in the study;
* If it is discovered that you do not meet the study requirements;
* If the study is canceled; or
* For administrative reasons.

If you leave the study for any reason, the study doctor may ask you to have some end-of-study tests for your safety.

Acknowledgment and Consent

The purpose, goals, expectations and risks of this study have been adequately explained to me. I hereby give my consent to be enrolled. I understand that enrollment is completely voluntary and that no proven available treatment will be withheld from me if I decided not to enroll in the study. I understand that I may withdraw from participation this study at any time without any penalty. I understand that my authorization and consent to use my information expires at the end of this research study. The information gathered from this study is considered protected health information and that information which is presented in scientific meetings or published in the medical literature will not include my name or any information that identifies me to anyone hearing or reading the report.

_________________________ Subject's Printed Name

* _________________________ _________________________ Subject's Signature Date

Printed Name of Person Conducting the Consent Discussion

_________________________ _________________________ Signature of the Person Conducting Date the Consent Discussion

AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

If you decide to be in this study, the study doctor and study staff will use and share health data about you to conduct the study. Health data may include:

* Your name.
* Address.
* Phone number.
* Date of birth.
* Medical history.
* Information from your study visits, including all test results.

Health data may come from your study records or from existing records kept by your doctor or other health care workers.

For this study, the study staff may share health data about you with authorized users. Authorized users may include:

* Representatives of Helm Vision Group.
* Representatives of Advarra IRB (an Institutional Review Board that reviews this study).
* The Food and Drug Administration (FDA) and other US federal and state agencies.
* Government agencies to whom certain diseases (like HIV, hepatitis, and STDs) must be reported.
* Governmental agencies of other countries.
* Outside individuals and companies, such as laboratories and data storage companies, that work with the researchers and sponsor and need to access your information to conduct this study.
* Other research doctors and medical centers participating in this study, if applicable.
* A data safety monitoring board which oversees this study, if applicable.

Your health data will be used to conduct and oversee the research, including for instance:

* To see if the study treatment works and is safe.
* To compare the study treatment to other treatments.
* For other research activities related to the study treatment.

Once your health data has been shared with authorized users, it may no longer be protected by federal privacy law and could possibly be used or disclosed in ways other than those listed here.

Your permission to use and share health data about you will end in 50 years unless you revoke it (take it back) sooner.

You may revoke (take back) your permission to use and share health data about you at any time by writing to the study doctor at the address listed on the first page of this form. If you do this, you will not be able to stay in this study. No new health data that identifies you will be gathered after your written request is received. However, health data about you that has already been gathered may still be used and given to others as described in this form.

Your right to access your health data in the study records will be suspended during the study to keep from changing the study results. When the study is over, you can access your study health data.

If you decide not to sign and date this form, you will not be able to take part in the study.

STATEMENT OF AUTHORIZATION I have read this form and its contents were explained. My questions have been answered. I voluntarily agree to allow study staff to collect, use and share my health data as specified in this form. I will receive a signed and dated copy of this form for my records. I am not giving up any of my legal rights by signing and dating this form.

_________________________ Subject's Printed Name

_________________________ _________________________ Subject's Signature Date

ELIGIBILITY:
Inclusion Criteria:Voluntary participation of subjects with moderate to dense sleeves with no allergy to ivermectin and the ability to keep follow-up appointments.

-

Exclusion Criteria: Patients under 18 years old and those allergic to ivermectin.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparative density of sleeves | Each patient will be followed for 6 months.
  The density of sleeves will be clinically assessed and graded by the outcomes assessor

SECONDARY OUTCOMES:
Comparative assessment of tear osmolarity between treated and untreated eyes | Each patient will be followed for 6 months
  The tear osmolarity will be tested in each eye at each follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Helm Vision Group, Santa Clarita, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share data with other researchers, unless requested.

REFERENCES:
- [Result] Choi Y, Eom Y, Yoon EG, Song JS, Kim IH, Kim HM. Efficacy of Topical Ivermectin 1% in the Treatment of Demodex Blepharitis. Cornea. 2022 Apr 1;41(4):427-434. doi: 10.1097/ICO.0000000000002802. PMID 34173370